CLINICAL TRIAL: NCT01160276
Title: An Open Non Randomized Comparative Study Exploring Drug Interaction Between Colchicine and Calcineurin Inhibitors in 2 Groups (Ciclosporin Group and Tacrolimus Group) of Renal Graft Recipients
Brief Title: Drug Interaction Between Colchicine and Calcineurin Inhibitors in Renal Graft Recipients
Acronym: COLCHINCAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081105
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Renal Replacement Therapies
Keywords: renal graft; colchicine; drug interaction; cyclosporine; tacrolimus; renal transplantation; renal transplant; ABCB1; CYP3A5; SLCO1B1
MeSH Terms: interventions — Colchicine; colchimax; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine (Active Comparator): The first group is composed of 14 renal graft recipients under cyclosporine
  Interventions: Drug: cyclosporine+colchicine
- Tacrolimus (Active Comparator): The second group is composed of 14 renal graft recipients under tacrolimus
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: cyclosporine+colchicine — the 14 patients of the 1st group are under cyclosporine and One pill of colchimax 1mg will be taken by all the patients at Day 3.
  Other Names: Colchicine; Colchimax
  Arms: Cyclosporine
Drug: tacrolimus — the 14 patients of the second group are under tacrolimus and One pill of colchimax 1mg will be taken by all the patients at Day 3.
  Other Names: Colchicine; Colchimax
  Arms: Tacrolimus

SUMMARY:
Ciclosporin inhibits P-glycoprotein should increase colchicine bioavailability whereas tacrolimus should not influence colchicine disposition.

This is a prospective, controlled, open labeled study performed in renal graft recipients comparing colchicine single dose (1mg) pharmacokinetics in 14 patients treated with tacrolimus and 14 patients treated with cyclosporin.

DETAILED DESCRIPTION:
* Renal transplantation >= one year
* eGFR (MDRD) > 30ml/min
* hemoglobin >= 11g/dl
* treatment with tacrolimus or cyclosporine
* no previous muscular disease
* no drugs interfering with P-glycoprotein or CYP3A activity or expression outcomes
* colchicine AUC, Cmax, T1/2
* ABCB1C3435T, CYP3A5 and SLCO1B1 genotypes

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal graft since at least 1 year
* Patients treated with ciclosporin or tacrolimus
* Are at least 18 years old.
* Glomerular filtration rate above 30 ml / min calculated using the MDRD formula
* Among the 14 patients receiving ciclosporin:
* The genotype is not a criterion for inclusion
* Among the 14 patients with tacrolimus treatment:
* 7 genotype ABCB1 3435CC, 7 genotype ABCB1 3435TT
* Recent (1 month) residual concentration of tacrolimus between 5-10ng/ml
* Recent (1 month) residual concentration of ciclosporin between 100-200ng/ml
* For women : a negative pregnancy test (serum beta hCG)
* Realization of a medical examination.
* Informed consent and writing form.

Exclusion Criteria:

* Abnormal transaminases (AST and ALT above the ULN Laboratory).
* Underlying Liver Disease (steatosis, cirrhosis, chronic hepatitis, the virus of hepatitis C or B).
* Previous history of muscle disease (drug related especially the statin type).
* Leukopenia (WBC <3000/mm3).
* Hemoglobin <11g/dl.
* Patient treated by erythropoetin (whatever its hemoglobin value).
* Abnormal CPK (greater than the ULN Laboratory).
* Prior intolerance to colchicine.
* Regular intake of the following medications associated with rhabdomyolyses: antipsychotics, cholesterol lowering agents (statins or fibrates), zidovudine, antidepressants (selective inhibitor of serotonin reuptake) and lithium.
* Patient (e) can not refrain from consuming grapefruit juice.
* Patient (e) taking a tea based on St John's wort.
* Taking drugs inducers of P-gp or CYP3A4 (rifabutin, rifampin, carbamazepine, phenytoin, phenobarbital, efavirenz, nevirapine, protease inhibitors, griseofulvin).
* Taking drugs inhibitors of P-gp or CYP3A4 (quinidine, macrolide antibiotics, azole antifungals, protease inhibitors, amiodarone, diltiazem, verapamil).
* Chronic diarrhea.
* ABCB1 Genotype 3435CT for patients in the tacrolimus group.
* Participation in another concurrent trial.
* Patient (e) exclusion period of another trial.
* Patient (e) having reached the maximum annual amount of compensation provided by law.
* No affiliation to French social security scheme or without CMU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve of plasma concentration of colchicine over time 0-∞ | 4 weeks

SECONDARY OUTCOMES:
Half-life of colchicine (T1/2). | 4 weeks
AUC0-3h colchicine to focus the analysis on the absorption phase (argument in favor of an interaction-dependent P-gp) | 4 weeks
Cmax observed colchicine. | 4 weeks
Residual tacrolimus or cyclosporine concentrations | 4 weeks
ABCB1 genotype at position 3435 (rs 1045642) or 3435 cc, 3435TT, heterozygotes could not be included in the tacrolimus group. | 4 weeks
ABCB1 Haplotypes composed of 3 SNPs: C3435T, G2677T / A and C1236T. | 4 weeks
CYP3A5 Genotype: search for the allele * 1 (rs 776746): 3 possible genotypes CYP3A5 * 3 / * 3 - CYP3A5 * 3 / * 1 - CYP3A5 * 1 / * 1. | 4 weeks
GFR calculated by MDRD formula. | 4 weeks
BMI | 4 weeks
Drug related (azathioprine, mycophenolic acid, diuretics, ACE inhibitors, ARAII) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Jacquet, MD, Principal Investigator — Nephrology Department of BICETRE Hospital
Locations (1):
- Assistance publique - Hôpitaux de Paris : Bicêtre Hospital, Le Kremlin-Bicêtre, France